CLINICAL TRIAL: NCT02043067
Title: Enhanced TB Screening to Determine the Prevalence and Incidence of TB in a Cohort of HIV Clinic Patients in Lusaka, Zambia
Brief Title: Enhanced TB Screening to Determine the Prevalence and Incidence of TB in Patients With HIV
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CIDRZ 1226/IRB12-0416
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2014-12

CONDITIONS: Tuberculosis
Keywords: TB; HIV; Extensively resistant TB; Extra pulmonary TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Additional samples (10 ml blood, and 20 ml urine) will be stored in the specimen repository at the CIDRZ laboratory for future studies. For patients who agree to provide samples for the repository and are diagnosed with TB, isolates from positive cultures (blood, urine, and/or sputum) will also be stored in the repository.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- new HIV clinic enrollees: All new enrollees to a Lusaka HIV clinic will receive a full TB work-up.
  Interventions: Other: Comprehensive TB screening

INTERVENTIONS:
Other: Comprehensive TB screening — All enrollees will receive a comprehensive TB screening regardless of symptom presentation.

SUMMARY:
This study will examine an enhanced protocol to systematically screen a cohort of 400 new HIV clinic enrollees for prevalence and 1-year incidence of tuberculosis (TB).

DETAILED DESCRIPTION:
Zambia is a high burden country for both HIV and TB infection and HIV clinic enrollees are a high-risk group for active TB. Current Zambian Ministry of Health screening protocols are symptom-based even though active case-finding studies in HIV-infected populations have shown that symptoms are not always predictive of active TB. As a result, there may be a significant amount of un-diagnosed TB among HIV-infected Zambians even in the context of accessing HIV care. This study will examine an enhanced protocol to systematically screen a cohort of 400 new HIV clinic enrollees for prevalence and 1-year incidence of TB using symptoms, light and fluorescence microscopy, chest radiography and TB culture of sputum and extra-pulmonary fluids (when indicated). In addition, the sensitivity, specificity and cost-effectiveness of each diagnostic tool will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Persons with HIV/AIDS, 16 years of age or older, who are enrolling at the Kalingalinga ART clinic and are able and willing to provide informed consent
* Antiretroviral therapy-naïve except for short-course therapy through prevention of mother-to-child-transmission programs
* Not have taken any TB treatment in the past 3 months
* Willing to provide locator information and allow study staff to contact by phone or visit them at home if required

Exclusion Criteria:

* Any condition, including active drug or alcohol use, which in the opinion of the investigators, would interfere with adherence to study requirements

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Four hundred new enrollees at the Kalingalinga HIV Care and Treatment Clinic who are not currently being treated for TB.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of undiagnosed TB in those with HIV. | Enrollment screening visit
  Among the cohort of 400 new enrollees at the clinic, all will be tested for TB at the specified time points using enhanced TB screening. Initial diagnosis will use smear microscopy and culture. Chest X-ray will be performed on the second day of enrollment. Presumptive Diagnosis: As culture results will take several days or weeks to become available, a presumptive diagnosis will be made based on history and physical exam, symptoms, smear microscopy and chest radiography results. All patients who are smear-positive by at least one sample will be diagnosed with TB per national guidelines. Patients who are smear-negative or suspected of extra-pulmonary TB based on clinical or radiographic findings may be treated empirically for TB at the discretion of a clinical or medical officer. Sputum samples will also be sent for testing at the end of the study with the Xpert MTB/RIF assay.

SECONDARY OUTCOMES:
Incidence of TB in a cohort of HIV clinic patients screened as 'TB negative'. | enrollment, 3, 6, 9 and 12 month visits.
  To account for patients who are censored prior to 12 months of follow-up, the incidence of TB will be calculated as a rate. Each patient will contribute follow-up time until they are censored, are diagnosed with TB, or have been in the study for 12 months. Patients who were diagnosed with TB at enrollment will not be included.

OTHER OUTCOMES:
Performance of diagnostic measures | Days 1, 2, 3; Months 3, 6 9 and 12
  The performance of symptom screening, light microscopy, fluorescence microscopy, chest x-ray, and Xpert MTB/RIF assay compared to culture of sputum and other fluids in HIV-infected patients will be evaluated using data analysis methods.
Cost-effectiveness of each screening/diagnostic tool. | Days 1, 2, 3 and months 3, 6, 9 and 12
  The primary outcomes of each diagnostic tool (or combination of diagnostic tools) that will be assessed are: cost per case diagnosed/detected, cost per patient cured, cost per case averted. For instance, the cost per case of active TB detected using the "null" or gold standard screening option will be calculated and compared to the cost per case of active TB detected using each of the other screening options.
Clinical outcomes | up to 12 months post-enrollment
  Clinical outcomes will be measured in a cohort of HIV-infected patients and TB/HIV co-infected patients during the first 12 months of HIV care including but not limited to mortality, immune recovery and development of other opportunistic infections.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Reid, MD, Principal Investigator — CIDRZ; University of North Carolina at Chapel Hill
Locations (1):
- Kalingalinga HIV Care and Treatment Clinic, Lusaka, Zambia

REFERENCES:
- [Background] Harris JB, Hatwiinda SM, Randels KM, Chi BH, Kancheya NG, Jham MA, Samungole KV, Tambatamba BC, Cantrell RA, Levy JW, Kimerling ME, Reid SE. Early lessons from the integration of tuberculosis and HIV services in primary care centers in Lusaka, Zambia. Int J Tuberc Lung Dis. 2008 Jul;12(7):773-9. PMID 18544203
- [Background] Moore D, Liechty C, Ekwaru P, Were W, Mwima G, Solberg P, Rutherford G, Mermin J. Prevalence, incidence and mortality associated with tuberculosis in HIV-infected patients initiating antiretroviral therapy in rural Uganda. AIDS. 2007 Mar 30;21(6):713-9. doi: 10.1097/QAD.0b013e328013f632. PMID 17413692
- [Background] Mohammed A, Ehrlich R, Wood R, Cilliers F, Maartens G. Screening for tuberculosis in adults with advanced HIV infection prior to preventive therapy. Int J Tuberc Lung Dis. 2004 Jun;8(6):792-5. PMID 15182152
- [Background] Day JH, Charalambous S, Fielding KL, Hayes RJ, Churchyard GJ, Grant AD. Screening for tuberculosis prior to isoniazid preventive therapy among HIV-infected gold miners in South Africa. Int J Tuberc Lung Dis. 2006 May;10(5):523-9. PMID 16704034
- [Background] Lawn SD, Myer L, Bekker LG, Wood R. Burden of tuberculosis in an antiretroviral treatment programme in sub-Saharan Africa: impact on treatment outcomes and implications for tuberculosis control. AIDS. 2006 Aug 1;20(12):1605-12. doi: 10.1097/01.aids.0000238406.93249.cd. PMID 16868441
- [Background] Wood R, Middelkoop K, Myer L, Grant AD, Whitelaw A, Lawn SD, Kaplan G, Huebner R, McIntyre J, Bekker LG. Undiagnosed tuberculosis in a community with high HIV prevalence: implications for tuberculosis control. Am J Respir Crit Care Med. 2007 Jan 1;175(1):87-93. doi: 10.1164/rccm.200606-759OC. Epub 2006 Sep 14. PMID 16973982
- [Background] Wise J. Southern Africa is moving swiftly to combat the threat of XDR-TB. Bull World Health Organ. 2006 Dec;84(12):924-5. No abstract available. PMID 17242824
- [Background] Behr MA, Warren SA, Salamon H, Hopewell PC, Ponce de Leon A, Daley CL, Small PM. Transmission of Mycobacterium tuberculosis from patients smear-negative for acid-fast bacilli. Lancet. 1999 Feb 6;353(9151):444-9. doi: 10.1016/s0140-6736(98)03406-0. PMID 9989714
- [Background] Hernandez-Garduno E, Cook V, Kunimoto D, Elwood RK, Black WA, FitzGerald JM. Transmission of tuberculosis from smear negative patients: a molecular epidemiology study. Thorax. 2004 Apr;59(4):286-90. doi: 10.1136/thx.2003.011759. PMID 15047946
- [Background] Kimerling ME, Schuchter J, Chanthol E, Kunthy T, Stuer F, Glaziou P, Ee O. Prevalence of pulmonary tuberculosis among HIV-infected persons in a home care program in Phnom Penh, Cambodia. Int J Tuberc Lung Dis. 2002 Nov;6(11):988-94. PMID 12475145
- [Background] Ba F, Rieder HL. A comparison of fluorescence microscopy with the Ziehl-Neelsen technique in the examination of sputum for acid-fast bacilli. Int J Tuberc Lung Dis. 1999 Dec;3(12):1101-5. PMID 10599014
- [Background] Mugusi F, Villamor E, Urassa W, Saathoff E, Bosch RJ, Fawzi WW. HIV co-infection, CD4 cell counts and clinical correlates of bacillary density in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2006 Jun;10(6):663-9. PMID 16776454
- [Background] Siddiqi K, Lambert ML, Walley J. Clinical diagnosis of smear-negative pulmonary tuberculosis in low-income countries: the current evidence. Lancet Infect Dis. 2003 May;3(5):288-96. doi: 10.1016/s1473-3099(03)00609-1. PMID 12726978
- [Background] Bakari M, Arbeit RD, Mtei L, Lyimo J, Waddell R, Matee M, Cole BF, Tvaroha S, Horsburgh CR, Soini H, Pallangyo K, von Reyn CF. Basis for treatment of tuberculosis among HIV-infected patients in Tanzania: the role of chest x-ray and sputum culture. BMC Infect Dis. 2008 Mar 6;8:32. doi: 10.1186/1471-2334-8-32. PMID 18325120
- [Background] Swaminathan S, Paramasivan CN, Kumar SR, Mohan V, Venkatesan P. Unrecognised tuberculosis in HIV-infected patients: sputum culture is a useful tool. Int J Tuberc Lung Dis. 2004 Jul;8(7):896-8. PMID 15260283
- [Background] Stringer JS, Zulu I, Levy J, Stringer EM, Mwango A, Chi BH, Mtonga V, Reid S, Cantrell RA, Bulterys M, Saag MS, Marlink RG, Mwinga A, Ellerbrock TV, Sinkala M. Rapid scale-up of antiretroviral therapy at primary care sites in Zambia: feasibility and early outcomes. JAMA. 2006 Aug 16;296(7):782-93. doi: 10.1001/jama.296.7.782. PMID 16905784
- [Background] Steingart KR, Henry M, Ng V, Hopewell PC, Ramsay A, Cunningham J, Urbanczik R, Perkins M, Aziz MA, Pai M. Fluorescence versus conventional sputum smear microscopy for tuberculosis: a systematic review. Lancet Infect Dis. 2006 Sep;6(9):570-81. doi: 10.1016/S1473-3099(06)70578-3. PMID 16931408
- [Background] Ministry of Health, Human Resources for Health: Strategic Plan 2006-2010. Ministry of Health, Ndeke House, Lusaka. 2006.
- [Background] Boehme CC, Nicol MP, Nabeta P, Michael JS, Gotuzzo E, Tahirli R, Gler MT, Blakemore R, Worodria W, Gray C, Huang L, Caceres T, Mehdiyev R, Raymond L, Whitelaw A, Sagadevan K, Alexander H, Albert H, Cobelens F, Cox H, Alland D, Perkins MD. Feasibility, diagnostic accuracy, and effectiveness of decentralised use of the Xpert MTB/RIF test for diagnosis of tuberculosis and multidrug resistance: a multicentre implementation study. Lancet. 2011 Apr 30;377(9776):1495-505. doi: 10.1016/S0140-6736(11)60438-8. Epub 2011 Apr 18. PMID 21507477
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Theron G, Peter J, van Zyl-Smit R, Mishra H, Streicher E, Murray S, Dawson R, Whitelaw A, Hoelscher M, Sharma S, Pai M, Warren R, Dheda K. Evaluation of the Xpert MTB/RIF assay for the diagnosis of pulmonary tuberculosis in a high HIV prevalence setting. Am J Respir Crit Care Med. 2011 Jul 1;184(1):132-40. doi: 10.1164/rccm.201101-0056OC. Epub 2011 Apr 14. PMID 21493734
- [Background] Lawn SD, Bekker LG, Miller RF. Immune reconstitution disease associated with mycobacterial infections in HIV-infected individuals receiving antiretrovirals. Lancet Infect Dis. 2005 Jun;5(6):361-73. doi: 10.1016/S1473-3099(05)70140-7. PMID 15919622
- [Background] Colebunders R, John L, Huyst V, Kambugu A, Scano F, Lynen L. Tuberculosis immune reconstitution inflammatory syndrome in countries with limited resources. Int J Tuberc Lung Dis. 2006 Sep;10(9):946-53. PMID 16964782
- [Background] Lawn SD, Wilkinson RJ, Lipman MC, Wood R. Immune reconstitution and "unmasking" of tuberculosis during antiretroviral therapy. Am J Respir Crit Care Med. 2008 Apr 1;177(7):680-5. doi: 10.1164/rccm.200709-1311PP. Epub 2008 Jan 17. PMID 18202347
- [Background] Meintjes G, Lawn SD, Scano F, Maartens G, French MA, Worodria W, Elliott JH, Murdoch D, Wilkinson RJ, Seyler C, John L, van der Loeff MS, Reiss P, Lynen L, Janoff EN, Gilks C, Colebunders R; International Network for the Study of HIV-associated IRIS. Tuberculosis-associated immune reconstitution inflammatory syndrome: case definitions for use in resource-limited settings. Lancet Infect Dis. 2008 Aug;8(8):516-23. doi: 10.1016/S1473-3099(08)70184-1. PMID 18652998
- [Background] Francis J. Curry National Tuberculosis Center Institutional Consultation Services, Conducting Sputum Induction Safely. 1999.
- [Background] Dasgupta K, Menzies D. Cost-effectiveness of tuberculosis control strategies among immigrants and refugees. Eur Respir J. 2005 Jun;25(6):1107-16. doi: 10.1183/09031936.05.00074004. PMID 15929967
- See also: University of North Carolina website — http://www.unc.edu